CLINICAL TRIAL: NCT04882215
Title: Development and Evaluation of a Novel Treatment Intervention for People With Acquired Brain Injury
Brief Title: Integrated PRocess and StrategieS Training: I-PRESS Training
Acronym: I-PRESS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to secure further funding to resume study activities.
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: GN19NE479
Record Dates: First submitted 2021-04-26; First posted 2021-05-11 (Actual); Results first posted 2024-11-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2023-11

CONDITIONS: Acquired Brain Injury
Keywords: Traumatic Brain Injury; Stroke; executive dysfunction
MeSH Terms: conditions — Brain Injuries; Brain Injuries, Traumatic; Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adaptive Training (AT) (Experimental): For AT participants, difficulty of the training tasks is progressively increased in response to task performance.
  Interventions: Behavioral: GMT combined with WMU Training
- Non Adaptive Training (NA) (Active Comparator): For NA participants, task difficulty is fixed at a relatively low level across all sessions.
  Interventions: Behavioral: GMT combined with WMU Training

INTERVENTIONS:
Behavioral: GMT combined with WMU Training — GMT teaches the use of mental strategies to support sustained attention during complex (multi-step) task performance following an interactive programme. GMT is structured into nine modules, with interactive discussions and homework assignments. It will be conducted on a group basis.
  WMU training consists of computerised working memory updating tasks in which trial accuracy and response time are recorded. Two tasks will be trained: 1. a visuo-spatial Matrix Updating (MU) and 2. a verbal Keep Track (KT). For both training tasks, level of difficulty can be modulated by increasing or decreasing the update level, i.e., the number of updates on each trial.

SUMMARY:
There is a pressing need to develop more effective interventions to remediate cognitive deficits in highly prevalent disabling conditions such as stroke, head injury and other forms of acquired brain injury (ABI). Neuropsychological rehabilitation interventions developed in a clinical setting have shown some beneficial effects, but the effectiveness of clinical interventions have potential to be enhanced if informed by findings from cognitive neuroscience. Research into cognitive training using methods such as functional magnetic resonance imaging (fMRI) has contributed to an understanding of factors that promote changes in brain function, but this approach seldom includes individuals with brain damage or cognitive deficits. Its potential for application with clinical populations is therefore uncertain, meaning that people who may benefit do not have access to interventions that may improve their health and wellbeing.

The proposed research brings together methods from neuropsychological rehabilitation and cognitive neuroscience to investigate 1) the feasibility of, and effect sizes arising from, combining an existing clinical intervention targeting mental strategies with an adaptive training programme targeting core cognitive processes, and 2) whether the novel treatment combination promotes changes in brain function that are detectable using fMRI.

This project will develop and evaluate a training intervention that aims to improve outcomes from a strategy-based rehabilitation intervention, Goal Management Training (GMT), by adding process-based cognitive training with adaptive difficulty to enhance the executive function of working memory updating (WMU). People with ABI (n=32) will complete 9 sessions of GMT, a recommended treatment for deficits in frontal-lobe executive functions, with the addition of 8 WMU training sessions with or without adaptive training. Measures of feasibility, acceptability, and fidelity will be taken, and effect sizes of differences in pre- to post-training changes on neural, cognitive, and functional measurements will be determined by comparing two experimental groups in which difficulty of the WMU training tasks either adaptively increases in response to performance or is fixed.

DETAILED DESCRIPTION:
Globally, stroke and head injury are leading causes of disability. Deficits in cognitive functions are common in these conditions, including impairment in frontal-lobe 'executive' functions such as working memory and the ability to solve problems, plan, and regulate actions in order to achieve intended goals. These deficits affect individuals' ability to live independently, work, and maintain social relationships. We propose that improving outcomes for people with acquired brain injury (ABI) requires an interdisciplinary approach in which neuropsychological rehabilitation and cognitive neuroscience complement one another.

In neuropsychological rehabilitation, interventions are classified as 'restorative' (restoration of underlying core cognitive processes including executive functions) or 'compensatory' (compensation of function through the use of external aids or learned strategies). Clinical guidelines recommend the use of 'meta-cognitive strategy training' for the treatment of deficits in frontal-lobe executive functions. Goal Management Training (GMT) is one such validated meta-cognitive strategy. GMT trains compensatory mental strategies to manage attention during multi-step tasks. GMT has been evaluated behaviourally in randomised controlled trials with positive, albeit modest, outcomes in individuals with ABI.

In cognitive neuroscience, an emerging research area concerns experience-induced neural changes referred to as neural plasticity. These may involve neural changes in: 1) task-based functional activation patterns, i.e. activity increases, decreases, or reorganisation, 2) brain structure, i.e., grey matter and white matter volume changes and 3) functional connectivity, i.e. changes in connectivity between brain regions that are recruited for a mental procedure as well as changes in the strength and magnitude.

Neuroimaging studies have demonstrated that programmes to train core cognitive processes including working memory (WM) executive functions can drive changes both in behavioural and neural measures. Performance gains after process-based training have been observed by several authors employing different training tasks and including both younger and older populations. In addition, generalisation to broad cognitive abilities such as reasoning, episodic memory, after process-based training, has been observed in both young and older adults although this area is under debate. This work has primarily involved healthy adults and whether the same findings apply to those with ABI needs to be investigated.

This research study aims to develop and evaluate a novel treatment intervention for people with ABI that combines a process-based cognitive training with a strategy-based GMT rehabilitation intervention, and to acquire functional magnetic resonance imaging (fMRI) data before and after the intervention to measure patterns of brain activity associated with a task requiring executive functions. We propose that outcomes from GMT might be improved by an adaptive, process-based intervention aimed at enhancing working memory processes. Adaptive task difficulty involves dynamic adjustment of training task demands so that the individual remains within an optimal range of performance.

i. Aims

The primary aim of the study is to investigate whether it is feasible and acceptable to deliver a novel intervention combining GMT with WMU training, within a randomised controlled trial (RCT) context in a sample of ABI individuals. A further aim is to examine the behavioural and neural changes related to the novel intervention as well as the effect sizes.

ii. Research Question

This project will combine methods from neuropsychological rehabilitation and cognitive neuroscience to answer the following: 1) Is it feasible to combine an existing treatment for executive dysfunction, GMT, with an adaptive WMU training and how much benefit is gained? 2) Does the novel treatment combination promote neural plasticity that is detectable using fMRI?

iii. Outcomes

Primary outcomes will be measures of feasibility, acceptability, and fidelity.

Secondary outcomes will be pre- to post-training change in behavioural data (i.e., neuro-psychological assessment battery, measures of cognitive task performance and everyday functioning) and fMRI data (i.e., task-related brain activity), analysed by training condition. In addition, exploratory analyses of individual differences in responsiveness to WMU training will be performed, by calculating correlations between amount of adaptive training task improvement and pre- to post-training change on neural, cognitive, and functional measurements.

iv. Design

Randomised controlled trial methodology; specifically stratified randomisation in conjunction with permuted block random allocation, using an active control group will compare two conditions: (1) GMT combined with adaptive training [AT]; (2) GMT combined with non-adaptive [NA] training. Thirty-two adults with non-progressive ABI sustained in adulthood will be recruited from the NHS.. Participants will complete a combination of standard GMT (9 sessions) and 8 WMU (AT or NA) training sessions, delivered in small groups. Neuropsychological and functional assessments will be performed before and after the intervention. In addition, fMRI scanning sessions will be conducted pre- and post-training

ELIGIBILITY:
Inclusion Criteria:

* Only those able to give informed consent and able to comply with the training protocol will be included.
* ≥ 6 months post-ABI at time of recruitment (expression of interest to participate either verbally or in writing)
* Adults over the age of 18.
* English language fluency (speaking)
* a combination of self/relative/friend/carer reports of everyday organisation/memory problems

Exclusion Criteria:

* Individuals with contra-indications to MRI (e.g. heart pacemaker)
* Comorbid progressive neurological disorder or neurodegenerative condition (e.g. dementia)
* Major psychiatric disorder considered likely to prevent engagement in the intervention programme (pre-ABI history of mood disorder or stable antidepressant medication will not lead to exclusion)
* History of major substance abuse problems likely to prevent engagement in the intervention programme
* Unable to give informed consent
* Unable to cooperate with the study protocol (e.g. severe impairment of hearing, vision or language)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-05-18 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2023-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Evans, PhD, DClin, Principal Investigator — University of Glasgow
Locations (1):
- Lead Communirty Brain Injury Team NHS Lanarkshire Law House Airdrie Road, Carluke, Lanarkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cicerone KD, Langenbahn DM, Braden C, Malec JF, Kalmar K, Fraas M, Felicetti T, Laatsch L, Harley JP, Bergquist T, Azulay J, Cantor J, Ashman T. Evidence-based cognitive rehabilitation: updated review of the literature from 2003 through 2008. Arch Phys Med Rehabil. 2011 Apr;92(4):519-30. doi: 10.1016/j.apmr.2010.11.015. PMID 21440699
- [Background] Tornas S, Lovstad M, Solbakk AK, Evans J, Endestad T, Hol PK, Schanke AK, Stubberud J. Rehabilitation of Executive Functions in Patients with Chronic Acquired Brain Injury with Goal Management Training, External Cuing, and Emotional Regulation: A Randomized Controlled Trial. J Int Neuropsychol Soc. 2016 Apr;22(4):436-52. doi: 10.1017/S1355617715001344. Epub 2016 Jan 26. PMID 26812574
- [Background] Brehmer Y, Kalpouzos G, Wenger E, Lovden M. Plasticity of brain and cognition in older adults. Psychol Res. 2014 Nov;78(6):790-802. doi: 10.1007/s00426-014-0587-z. Epub 2014 Sep 28. PMID 25261907
- [Background] Constantinidis C, Klingberg T. The neuroscience of working memory capacity and training. Nat Rev Neurosci. 2016 Jul;17(7):438-49. doi: 10.1038/nrn.2016.43. Epub 2016 May 26. PMID 27225070
- [Background] Klingberg T. Training and plasticity of working memory. Trends Cogn Sci. 2010 Jul;14(7):317-24. doi: 10.1016/j.tics.2010.05.002. Epub 2010 Jun 16. PMID 20630350
- [Background] Westerberg H, Klingberg T. Changes in cortical activity after training of working memory--a single-subject analysis. Physiol Behav. 2007 Sep 10;92(1-2):186-92. doi: 10.1016/j.physbeh.2007.05.041. Epub 2007 May 21. PMID 17597168
- [Background] Dahlin E, Neely AS, Larsson A, Backman L, Nyberg L. Transfer of learning after updating training mediated by the striatum. Science. 2008 Jun 13;320(5882):1510-2. doi: 10.1126/science.1155466. PMID 18556560
- [Background] Dahlin E, Backman L, Neely AS, Nyberg L. Training of the executive component of working memory: subcortical areas mediate transfer effects. Restor Neurol Neurosci. 2009;27(5):405-19. doi: 10.3233/RNN-2009-0492. PMID 19847067
- [Background] Jaeggi SM, Buschkuehl M, Jonides J, Perrig WJ. Improving fluid intelligence with training on working memory. Proc Natl Acad Sci U S A. 2008 May 13;105(19):6829-33. doi: 10.1073/pnas.0801268105. Epub 2008 Apr 28. PMID 18443283
- [Background] Buschkuehl M, Hernandez-Garcia L, Jaeggi SM, Bernard JA, Jonides J. Neural effects of short-term training on working memory. Cogn Affect Behav Neurosci. 2014 Mar;14(1):147-60. doi: 10.3758/s13415-013-0244-9. PMID 24496717
- [Background] Melby-Lervag M, Hulme C. Is working memory training effective? A meta-analytic review. Dev Psychol. 2013 Feb;49(2):270-91. doi: 10.1037/a0028228. Epub 2012 May 21. PMID 22612437
- [Background] Hsu NS, Novick JM, Jaeggi SM. The development and malleability of executive control abilities. Front Behav Neurosci. 2014 Jun 24;8:221. doi: 10.3389/fnbeh.2014.00221. eCollection 2014. PMID 25071485
- [Background] Jolles DD, Grol MJ, Van Buchem MA, Rombouts SA, Crone EA. Practice effects in the brain: Changes in cerebral activation after working memory practice depend on task demands. Neuroimage. 2010 Aug 15;52(2):658-68. doi: 10.1016/j.neuroimage.2010.04.028. Epub 2010 Apr 23. PMID 20399274

RESULTS

PARTICIPANT FLOW:
Groups:
- Adaptive Training (AT): Participants in this group receive a combination of Goal Management Training (GMT) and computerised Working Memory Updating (WMU). For participants in the AT group, difficulty of the Working Memory Updating (WMU) training tasks is progressively increased in response to task performance.
- Non Adaptive Training (NA): Participants in this group receive a combination of Goal Management Training (GMT) and computerised Working Memory Updating (WMU). For participants in the NA group, difficulty of the Working Memory Updating (WMU) training tasks remains at a relatively low level throughout the training period.
Period: Overall Study
Arm/Group | Adaptive Training (AT) | Non Adaptive Training (NA)
Started | 14 | 0
Completed | 9 | 0
Not Completed | 5 | 0
Not completed — Withdrawal by Subject | 5 | 0

BASELINE CHARACTERISTICS:
Population: In the context of disruptions associated with COVID-19, a decision was made to focus on testing the feasibility of running the experimental condition (Adaptive training) initially and therefore no participant was assigned in the control group (Non-Adaptive training).
Groups:
- Adaptive Training (AT): Participants in this group receive a combination of Goal Management Training (GMT) and computerised Working Memory Updating (WMU). For participants in the AT group, difficulty of the WMU training tasks is progressively increased in response to task performance.
- Non-Adaptive Training (NA): Participants in this group receive a combination of Goal Management Training (GMT) and computerised Working Memory Updating (WMU). For participants in the NA group, difficulty of the WMU training tasks remains at a relatively low level throughout the training period.
- Total: Total of all reporting groups
Arm/Group | Adaptive Training (AT) | Non-Adaptive Training (NA) | Total
Number analyzed (Participants) | 14 | 0 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.14 (10.49) |  | 53.14 (10.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 |  | 7
  Male | 7 |  | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 14 |  | 14

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Recruitment Process.
Description: Number of people referred from NHS eligible for screening and those entering the intervention. This will be continuously monitored throughout the study period.
Time Frame: From pre-intervention (Week 1) to post-intervention (Week 12).
Population: as for baseline characteristics
Measure: Number; unit: % participants entered the intervention
Groups:
- Non Adaptive Training (NA): Participants in this group receive a combination of Goal Management Training (GMT) and computerised Working Memory Updating (WMU). For participants in the NA group, difficulty of the WMU training tasks remains at a relatively low level throughout the training period.
Arm/Group | Adaptive Training (AT) | Non Adaptive Training (NA)
Number analyzed (Participants) | 42 | 0
% participants entered the intervention | 33.33 |

2. Primary Outcome: Participants' Drop-out Rates
Description: Number of people completing the intervention to assess drop-out rates. This will be continuously monitored throughout the study period.
Time Frame: From pre-intervention (Week 1) to post-intervention (Week 12).
Population: as for baseline characteristics
Measure: Number; unit: % of participants who dropped out
Arm/Group | Adaptive Training (AT) | Non Adaptive Training (NA)
Number analyzed (Participants) | 14 | 0
% of participants who dropped out | 35.7 |

3. Primary Outcome: Participants' Coherence and Adherence to the Intervention.
Description: Mean percentage of working memory training sessions completed (a total of eight) were calculated across participants.
Time Frame: From pre-intervention (Week 1) to post-intervention (Week 12).
Population: From the N=14 people entering the AT group, N=5 dropped out and therefore we analysed data from the remaining N=9 individuals. In the context of disruptions associated with COVID-19, a decision was made to focus on testing the feasibility of running the experimental condition (Adaptive training) initially and therefore no participant was assigned in the control group (Non-Adaptive training).
Measure: Mean (Standard Deviation); unit: % of working memory sessions completed
Arm/Group | Adaptive Training (AT) | Non-Adaptive Training (NA)
Number analyzed (Participants) | 9 | 0
% of working memory sessions completed | 73.61 (19.2) |

4. Primary Outcome: Feedback Questionnaire
Description: Participant evaluation of the intervention using a study-specific questionnaire including eight 5-point Likert-scale agreement questions (scores of 1 to 5 with 1 being positive and 5 being negative). Mean feedback score was calculated across participants.
Time Frame: Post-intervention session (Week 12)
Population: From the N=14 people entering the AT group, a total of N=5 dropped out and therefore we analysed data from the remaining N=9 individuals. In the context of disruptions associated with COVID-19, a decision was made to focus on testing the feasibility of running the experimental condition (Adaptive training) initially and therefore no participant was assigned in the control group (Non-Adaptive training).
Measure: Mean (Standard Deviation); unit: Average feedback score
Arm/Group | Adaptive Training (AT) | Non-Adaptive Training (NA)
Number analyzed (Participants) | 9 | 0
Average feedback score | 1.25 (0.31) |

5. Secondary Outcome: Visuospatial Working Memory Using the Visuospatial Matrix Updating fMRI Task
Description: Performance in visuospatial working memory using the visuospatial Matrix Updating fMRI task. Accuracy is calculated as the proportion of correct responses at low and high difficulty task trials. Post-intervention session was used to calculate this measure.
Time Frame: Post-intervention session (week 12)
Population: From the N=14 people entering the AT group, a total of N=7 people took part in the fMRI session. In the context of disruptions associated with COVID-19, a decision was made to focus on testing the feasibility of running the experimental condition (Adaptive training) initially and therefore no participant was assigned in the control group (Non-Adaptive training).
Measure: Mean (Standard Deviation); unit: proportion of correct responses
Arm/Group | Adaptive Training (AT) | Non-Adaptive Training (NA)
Number analyzed (Participants) | 7 | 0
proportion of correct responses | 0.69 (0.25) |

6. Secondary Outcome: Visuospatial Working Memory fMRI Task Accuracy Using the Spatial N-back fMRI Task
Description: Performance on spatial working memory using the spatial n-back fMRI task as calculated by proportion of correct responses at low and high difficulty n-back task trials. Post-intervention session was used to calculate this measure.
Time Frame: Post-intervention session (Week 12)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: proportion of correct responses
Arm/Group | Adaptive Training (AT) | Non-Adaptive Training (NA)
Number analyzed (Participants) | 7 | 0
proportion of correct responses | 0.78 (0.14) |

7. Secondary Outcome: Episodic Visual Memory Accuracy Using the Object-location Association fMRI Task.
Description: Performance on visual episodic memory using the Object-location association fMRI task calculated by the proportion of correct responses at low and high difficulty level task trials. Post-intervention session was used to calculate this measure.
Time Frame: Post-intervention session (Week 12)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: proportion of correct responses
Arm/Group | Adaptive Training (AT) | Non-Adaptive Training (NA)
Number analyzed (Participants) | 7 | 0
proportion of correct responses | 0.58 (0.15) |

8. Secondary Outcome: Changes in Shifting Attention Using the Intra-Extra Dimensional Set Shift Test Variant From CANTAB Connect Research Web-testing.
Description: Number of trials for which the outcome was an incorrect response (subject pressed the incorrect button within the response window), calculated across all assessed trials. Higher score indicates a worse outcome. Mean percentage change between pre and post intervention scores was calculated across participants.
Time Frame: Pre-intervention (Week 1) and post-intervention (Week 12)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: % change between pre and post scores
Arm/Group | Adaptive Training (AT) | Non-Adaptive Training (NA)
Number analyzed (Participants) | 9 | 0
% change between pre and post scores | 10.11 (80) |

9. Secondary Outcome: Changes in Spatial Planning and Problem Solving Using the Stockings of Cambridge Test Variant From CANTAB Connect Research Web-testing.
Description: Number of assessed problems that the participant successfully completed in the minimum possible number of moves. Calculated over all assessed trials. Higher score indicates a better outcome. Mean percentage change between pre and post intervention scores was calculated across participants.
Time Frame: Pre-intervention (Week 1) and post-intervention (Week 12)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: % change between pre and post scores
Arm/Group | Adaptive Training (AT) | Non-Adaptive Training (NA)
Number analyzed (Participants) | 9 | 0
% change between pre and post scores | 6.33 (30.75) |

10. Secondary Outcome: Changes in Spatial Working Memory Using the Spatial Working Memory Test Variant From CANTAB Connect Research Web-testing.
Description: The number of times the subject incorrectly revisits a box in which a token has previously been found. Calculated across all assessed four, six and eight token trials. Higher score indicates a worse outcome. Mean percentage change between pre and post intervention scores was calculated across participants.
Time Frame: Pre-intervention (Week 1) and post-intervention (Week 12)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: % change between pre and post scores
Arm/Group | Adaptive Training (AT) | Non-Adaptive Training (NA)
Number analyzed (Participants) | 9 | 0
% change between pre and post scores | 19.72 (48.64) |

11. Secondary Outcome: Changes in Visuospatial Working Memory Using the Spatial Span Forward Test Variant From CANTAB Connect Research Web-testing.
Description: The Spatial Span forward test variant from CANTAB connect research web-testing was used calculated by the longest sequence of boxes successfully recalled by the participant. Higher score indicates a better outcome. Mean percentage change between pre and post intervention scores was calculated across participants.
Time Frame: Pre-intervention (Week 1) and post-intervention (Week 12)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: % change between pre and post scores
Arm/Group | Adaptive Training (AT) | Non-Adaptive Training (NA)
Number analyzed (Participants) | 9 | 0
% change between pre and post scores | 3.70 (18.22) |

12. Secondary Outcome: Changes in Visuospatial Working Memory Using the Spatial Span Reverse Test Variant From CANTAB Connect Research Web-testing.
Description: The Spatial Span reverse test variant from CANTAB connect research web-testing was used calculated by the longest sequence of boxes successfully recalled. Higher score indicates a better outcome. Mean percentage change between pre and post intervention scores was calculated across participants.
Time Frame: Pre-intervention (Week 1) and Post-intervention (Week 12)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: % change between pre and post scores
Arm/Group | Adaptive Training (AT) | Non-Adaptive Training (NA)
Number analyzed (Participants) | 9 | 0
% change between pre and post scores | 14.89 (37.12) |

ADVERSE EVENTS:
Time Frame: Adverse data were collected for the duration of the study, i.e., for 12 weeks. That is from pre-intervention (Week 1) to post-intervention (Week 12).
Description: Safety Reporting for UK Health Departments' Research Ethics Service (RES):
  A serious adverse event (SAE) is defined as an untoward occurrence that:
  1. results in death;
  2. is life-threatening;
  3. requires hospitalisation or prolongation of existing hospitalisation;
  4. results in persistent or significant disability or incapacity; or
  5. consists of a congenital abnormality or birth defect; or
  6. is otherwise considered medically significant by the investigator.
Arm/Group | Adaptive Training (AT) | Non-Adaptive Training (NA)
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/0
Other Adverse Events (participants affected / at risk) | 0/14 | 0/0

LIMITATIONS AND CAVEATS:
The study was substantially disrupted by the COVID-19 pandemic. Due to this delay, the project funding supporting the researcher came to an end before finishing the study and therefore failed to hit the recruitment target. For this reason group analysis was not possible, therefore, the data were analysed on a case-study basis. Any group analysis should be interpreted with caution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-06): https://cdn.clinicaltrials.gov/large-docs/15/NCT04882215/Prot_SAP_000.pdf